CLINICAL TRIAL: NCT04448535
Title: Effects of Ginkgo (Gingko Biloba) on Retinal and Choroidal Ocular Tissue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York College of Optometry (Other)
Responsible Party: Principal Investigator, Alexandra Benavente, Associate Clinical Professor, State University of New York College of Optometry
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1619383-1
Record Dates: First submitted 2020-06-24; First posted 2020-06-26 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Healthy
MeSH Terms: interventions — Ginkgo Extract

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gingko Biloba (Experimental): oral intake of gingko biloba for 4 weeks
  Interventions: Dietary Supplement: Gingko Biloba

INTERVENTIONS:
Dietary Supplement: Gingko Biloba — oral intake of Gingko Biloba, 240mg/day for 4 weeks

SUMMARY:
The purpose of this study is to understand the effect of Ginkgo Biloba oral supplements on retinal and choroidal ocular tissue.

DETAILED DESCRIPTION:
The study objectives are to:

1. assess the changes from pre- to post- oral supplementation on retinal and choroidal thickness and blood flow, retinal oxygen saturation, ocular perfusion pressure, and retinal function

ELIGIBILITY:
Inclusion Criteria:

* Aged between 20 - 55 years, inclusive
* Good general and ocular health
* Corrected visual acuity of 20/40 or better
* No gingko biloba supplementation within the last 3 months

Exclusion Criteria:

* All significant ocular and any systemic disorders considered likely to affect the systemic or ocular vasculature
* History of ocular surgery, including refractive surgery
* Use of ocular medications
* Conditions where ginkgo supplementation is contraindicated
* Any eye or systemic disease that affect vision or refractive error
* Current smokers
* Subjects who are pregnant, breastfeeding, or planning conception

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2022-08-03 (Actual)

PRIMARY OUTCOMES:
ocular blood flow | 4 weeks
  ocular blood flow measured with doppler ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- SUNY College of Optometry, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No